CLINICAL TRIAL: NCT04752956
Title: Effectiveness of Sodium Hyaluronate In Relieving Nasal Symptoms Of Children With Seasonal Allergic Rhinitis
Acronym: EHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nazlı ERCAN, Pediatric Allergy and Immunology Specialist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA2021
Record Dates: First submitted 2021-01-31; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Grup1 (Active Comparator): Nasal steroid spray only (NS) (Each dose contains 27.5 micrograms of fluticasone furoate; administered single dose per day as 1 puff through both nostrils)
  Interventions: Other: "Total nasal symptom score" (TNSS); Behavioral: Paediatric Rhinoconjunctivitis Quality of Life Questionnaire" (PRQLQ); Diagnostic Test: Nasal cytology; Diagnostic Test: anterior rhinomanometry
- Grup 2 (Active Comparator): NS + administered ambient temperature normal saline (NSS) through both nostrils by means of nasal douche device twice a day 15 minutes before NS. (NSS; 0,09% NaCl, pH:4-5)
  Interventions: Other: "Total nasal symptom score" (TNSS); Behavioral: Paediatric Rhinoconjunctivitis Quality of Life Questionnaire" (PRQLQ); Diagnostic Test: Nasal cytology; Diagnostic Test: anterior rhinomanometry
- Grup 3 (Active Comparator): NS + administered ambient temperature hyaluronic acid (HA) through both nostrils by means of nasal douche device twice a day 15 minutes before NS. (Nasorinse plus pediatric® Ingredients: water, sodium chlorine, sodium bicarbonate, and HA; pH balanced)
  Interventions: Other: "Total nasal symptom score" (TNSS); Behavioral: Paediatric Rhinoconjunctivitis Quality of Life Questionnaire" (PRQLQ); Diagnostic Test: Nasal cytology; Diagnostic Test: anterior rhinomanometry

INTERVENTIONS:
Other: "Total nasal symptom score" (TNSS) — TNSS contains 4 parameters in assessing the severity of allergic rhinitis: nasal congestion, runny nose, nasal itching, and sneezing. Each symptom is scored out of 4 points, from 0 to 3. 0, none- there are no complaints 1- mild- any symptom that exists but is not particularly annoying; 2, moderate, - any annoying symptom but does not interfere with daily activities or sleep; 3, severe - any symptom preventing daily activities or disturbing during sleeping. The total score is calculated by summing all the scores of 4 fields, which vary ranges from 0 to 15 .In our study, all patients will be instructed to record their TNSS symptom scores on their diary cards each morning before taking the drug. Patients will be graded on baseline TNSS parameters compared to 4 weeks before starting treatment.
Behavioral: Paediatric Rhinoconjunctivitis Quality of Life Questionnaire" (PRQLQ) — PRQLQ, is a self-administered, disease-specific questionnaire, evaluating physical, emotional, and social status of individuals with AR. It contains 23 items in 5 domains: nose symptoms (RS), eye symptoms (ES), practical problems (PF), activity limitation (RL) and other symptoms (OS). One score is given to each domain. 7-point scale (from 0, not problematic; to 6, very problematic). The overall score is derived from the average score of all items (20). In our study, the Turkish validated form of PRQLQ was used
  Patients will be asked to answer PRQLQ questions at the end of each week during treatment. At the end of the treatment, an average of 4 weeks will be taken as the PRQLQ score. Basal PRQLQ questions will be evaluated by the participants based on 4 weeks prior to treatment.
Diagnostic Test: Nasal cytology — In anterior rhinoscopy, nasal cytology will be scraped off the middle part of the lower turbinate with the help of a small sterile cotton swab. The cellular material obtained will be fixed by air drying on a glass slide and then stained by the May-Grünwald-Giemsa method. Preparations that do not contain respiratory epithelium or contain less than 10 epithelium at high magnification will be excluded from the study. A percentage of cells per 100 cells will be reported. NECs (nasal eosinophilic count) will be evaluated according to the quantitative classification of Gelardi et al. An experienced cytologist who is blind to the study groups will perform this test. Eosinophil percentages in nasal smears of all patients will be evaluated before and after the treatment.
Diagnostic Test: anterior rhinomanometry — Children's right, left and total nasal airway resistance (NAR) and nasal airflow (NAF) will be measured with active anterior rhinomanometry ZAN 100 USB Rhinomanometry (Longmont, Colo., USA). In the evaluation, the NAR- pressure difference / air flow (R = P / V) formula will be used at a constant 150 Pascal prescribed by the European Rinomanometry Standardization Committee in 1984. After the patient is rested for 20 minutes, measurements will be made at 20-22 ° C and the nasal secretion will be cleared. NAR and NAF values of the participants will be measured before starting treatment and 4 weeks after treatment.

SUMMARY:
Nasal irrigation (NI) is recommended as an add-on therapy in patients with allergic rhinitis (AR). The primary purpose of this study was to evaluate the clinical effectiveness of adding hyaluronic acid (HA) solution and normal saline (NSS) to nasal steroid (NS) therapy as add - on therapy in improving quality of life and reducing nasal symptom scores of children with seasonal AR (SAR) with regards to NS therapy. Our secondary purpose was to demonstrate the effects on eosinophil count in nasal cytology (NEC), nasal airflow (NAF), and resistance (NAR).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 6 to 12-year-old;
* Children must have a clinical history concordant to seasonal allergic rhinitis of the previous year;
* Children must have skin prick test (SPT) positivity to pollen (tree, grass, or weed) (Positive SPT is defined as; skin reaction with within 15 minutes after the test and 3 mm larger swelling compared to the negative control test; ALK, Hørsholm, Denmark)
* Children must have a total nasal symptom score (TNSS) of 4 or more on 4 of 7 days during the run-in period.

Exclusion Criteria:

* Children who were treated with systemic/topical nasal corticosteroids, antihistamines or antibiotics, leukotriene receptor antagonists 4 weeks before the examination,
* those who had upper or lower respiratory tract infections;
* recipients of recent or ongoing allergen immunotherapy;
* active smokers;
* those with cystic fibrosis, immunodeficiency, septal deviation, nasal polyps, and ostio-metal complex, exudation, abnormal nasal diagnostic function, nasal anatomical disorder, metabolic disease, or congenital disease.
* Phone calls will measure children's adherence rate to treatment protocols, and participants determined to have treatment protocol adherence rates below 85% will be excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Estimated)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2021-06-06 (Estimated)

PRIMARY OUTCOMES:
Results of "total nasal symptom score" surveys | 28 days
  The primary outcome will be to understand whether nasal irrigation with hyaluronic acid (HA) solution will be beneficial as add-on therapy in children who are already receiving nasal steroid (NS) therapy.
  Total Nasal Symptom Scores (TNSS) of all participants (the study and control groups) will be used in grading the symptom relief of seasonal allergic rhinitis.
  Each symptom (nasal congestion, runny nose, nasal itching, and sneezing) will be graded from 0-3 (0=None, 1=Mild, 2=Moderate, 3=Severe) by the participants during the screening. No special unit for the scoring system is identified according to TNSS (Only scores mentioned with numbers will be analyzed with SPSS, and the percentages of symptoms will be the primary outcome).
Results of "Pediatric rhinoconjunctivitis quality of life questionnaire" survey | 28 days
  PRQLQ is a self-administered, disease-specific questionnaire and the survey contains 23 items in 5 domains: nose symptoms (RS), eye symptoms (ES), practical problems (PF), activity limitation (RL) and other symptoms (OS). One score is given to each domain. 7-point scale (from 0, not problematic; to 6, very problematic). The overall score will be derived from the average score of all items.
  No special unit for the scoring system is identified according to PRQLQ (Only scores mentioned with numbers will be analyzed with SPSS, and the percentages of symptoms will be the primary outcome 2).

SECONDARY OUTCOMES:
Nasal smear eosinophil count (percentages) | Two days
  • Nasal cytology in anterior rhinoscopy, the middle part of the lower concave will be scraped with the help of a small sterile cotton swab. Slides will be first screened under microscopes to determine the adequacy and cellular areas of the sample at 100 magnification. Slides will be dripped immersion oil and screened under an optic microscope x 1.000 magnification equipped with a digital camera. Analysis of rhino cystograms will involve screening at least 50 fields (300 cells). A percentage of the cell per 100 cells will be reported. NECs (nasal eosinophilic count) will be evaluated according to quantitative classification system described previously by Gelardi et al. Grade 0: No cell; Grade ½: 0,1-1% Eosinophil; Grade 1: 1.1-5% Eosinophil; Grade 2: 5-15% Eosinophil; Grade 3: 15-20% Eosinophil; Grade 4: > 20% Eosinophil. Eosinophil percentages in nasal smears of all patients will be evaluated before and at the end of treatment.
Nasal airflow (NAF) (ccm/sn) | Two days
  Nasal airflow (NAF) will be measured by means of active anterior rhinomanometry ZAN 100 USB Rhinomanometry (Longmont, Colo., USA) device. Measurements will be conducted at 20-22 °C after the patient rests for 20 minutes and the nasal secretion will be cleaned. NAF values of the participants will be measured before initiating the treatment and after 4 weeks of the treatment.
Nasal resistance (NAR) (Pa. s/ml) | Two days
  Nasal resistance (NAR) will be measured with active anterior rhinomanometry ZAN 100 USB Rhinomanometry device (Longmont, Colo., USA). In the evaluation, the formula NAR- pressure difference/airflow (R = P/V) will be used in the constant 150 Pascal stipulated by the European Rhinomanometry Standardization Committee in 1984.

CONTACTS AND LOCATIONS:
Overall Officials: Nazli Ercan, MD, Study Director — University of Health Sciences, Gulhane Research and Training Hospital, Department of Pediatrics
Locations (2):
- Turkey (Türkiye) (2):
  - Health Sciences University, Gülhane Training and Research Hospital, Gn. Dr. Tevfik Sağlam Cd No:11, Ankara, Etlik
  - Gülhane Training and Research Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Savietto E, Marioni G, Maculan P, Pettorelli A, Scarpa B, Simoni E, Astolfi L, Marchese-Ragona R, Ottaviano G. Effectiveness of micronized nasal irrigations with hyaluronic acid/isotonic saline solution in non-polipoid chronic rhinosinusitis: A prospective, randomized, double-blind, controlled study. Am J Otolaryngol. 2020 Jul-Aug;41(4):102502. doi: 10.1016/j.amjoto.2020.102502. Epub 2020 May 7. PMID 32460989
- [Derived] Ercan N, Demirel F, Yesillik S, Bolat A, Kartal O. Efficacy of sodium hyaluronate in relieving nasal symptoms of children with intermittent allergic rhinitis: a randomized controlled trial. Eur Arch Otorhinolaryngol. 2022 Jun;279(6):2925-2934. doi: 10.1007/s00405-021-07073-0. Epub 2021 Sep 16. PMID 34529156